CLINICAL TRIAL: NCT06721949
Title: Taurine Supplementation as a Novel Therapeutic Approach for Neurocognitive Symptoms in Long COVID
Brief Title: Taurine Supplementation in Long COVID
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RECLAIM -TaurineLC
Record Dates: First submitted 2024-11-28; First posted 2024-12-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Long COVID
Keywords: Taurine; COVID; Long COVID; randomized trial; neurocognitive symptoms
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Taurine

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taurine (Experimental): Participants randomized to the Taurine arm will receive two 675 mg taurine capsules twice daily for 12 weeks.
  Interventions: Drug: Taurine
- Placebo (Placebo Comparator): Participants randomized to the Placebo arm will receive two placebo capsules twice daily for 12 weeks. The placebo capsules will be visually identical to the taurine capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Taurine — Taurine is a naturally occurring amino sulfonic acid commonly found in the body. It is marketed as a natural health product/supplement and plays an important role in the body.
  Arms: Taurine
Drug: Placebo — The placebo capsule is visually identical to the taurine capsule.
  Arms: Placebo

SUMMARY:
The COVID-19 pandemic has swept across the globe, affecting millions of individuals with varying degrees of severity. While many individuals recover from the acute phase of the infection, a significant proportion continue to experience persistent and debilitating symptoms long after the initial SARS-CoV-2 infection. This condition, known as Long COVID (LC) or sometimes referred to as Post-COVID Condition (PCC) or post-acute sequelae of COVID-19, has emerged as a complex multisystemic condition and challenging health issue, affecting approximately 10% of COVID-19 patients. Various symptoms characterize LC, including fatigue, sleep disturbances, cognitive impairment, and mood disturbances. Some of the symptoms are shared with Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) - a condition marked by debilitating fatigue and a host of other symptoms without precise biomarkers or objective tests for diagnosis. Effective LC treatments remain elusive and LC patients continue to grapple with persistent symptoms that significantly impact their quality of life. Given the lack of effective treatments, it is imperative to explore novel therapeutic approaches that may alleviate the suffering of this patient population.

DETAILED DESCRIPTION:
Purpose: The overall trial objectives are to evaluate the efficacy and safety of taurine supplementation in treating and managing prolonged symptoms related to LC, focusing on neurocognitive-associated symptoms and fatigue.

Hypothesis: Increasing taurine levels in the body through treatment with taurine supplements will have a beneficial effect on Long COVID symptoms particularly neurocognitive-associated symptoms and fatigue.

Justification: Previous studies have suggested a correlation between low plasma taurine levels and symptoms associated with Long COVID. Reduced plasma taurine levels have also been observed in patients with Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS). The decreasing trajectory of taurine levels observed in long COVID could partly explain the fatigue, as taurine plays multiple roles in skeletal muscle function, the central nervous system, and energy metabolism. Furthermore, in various clinical and preclinical studies, including antioxidant, anti-aging, cytoprotective, and cardioprotective effects, taurine has demonstrated various therapeutic activities. Taurine also has a role in neuromodulation and the treatment of other central nervous system disorders, including depression. These findings suggest that taurine may be important in addressing the persistent symptoms and adverse outcomes in LC patients.

Given the robust association between taurine levels and symptoms and adverse outcomes of LC and the safety profile, there is a strong biological and clinical rationale for investigating taurine supplementation. There is a lack of effective treatments for LC, and exploring taurine supplementation as a novel therapeutic approach is justified and holds the potential to significantly improve the lives of affected individuals with an excellent safety profile.

Objectives: The overall trial objectives are to evaluate the efficacy and safety of taurine supplementation in treating and managing prolonged symptoms related to LC, focusing on neurocognitive-associated symptoms and fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Positive COVID-19 test by nasopharyngeal swab RT-PCR test, antibody or antigen tests at least 3 months prior to randomization; OR Presumed COVID-19 assessed by the site investigator (no positive COVID-19 test) with acute illness after October 15, 2019, and at least 3 months prior to randomization.
3. If participants have treatable symptoms, they should have had a stable regimen of treatment prior to entering the study (i.e. started treatment for at least 4 weeks).
4. Lingering COVID-19 symptoms beyond 3 months from onset of acute COVID and symptoms have lasted at least 2 months. The onset of COVID is considered the earliest of two dates: the date of positive testing or the date of first symptoms.
5. Lingering symptoms from COVID-19 present at the time of randomization.
6. Individuals of childbearing potential (as assessed by the overseeing Investigator) who are sexually active must agree to practice true abstinence or use at least one highly effective method of contraception while on study treatment. Highly effective methods of contraception must be discussed and approved by the overseeing Investigator (refer to Section 5 Contraception of the Master Protocol, and Section 13.1.2 of this protocol).
7. Must be able to provide informed consent and both willing and able to comply with study requirements.
8. Medications prescribed for treating fatigue or cognition have been discontinued for four weeks prior to enrolment and randomization. These include sildenafil, modafinil (Provigil), or armodafinil (Nuvigil), guanfacine, N-acetyl cysteine, and stimulant medications used for attention-deficit hyperactivity disorder (ADHD).

Exclusion Criteria:

1. Patients who had mechanical ventilation or extracorporeal membrane oxygen (ECMO) for COVID-19.
2. Current end-organ failure, organ transplantation, or current hospitalization in an acute care hospital.
3. Contraindications to the study intervention.
4. Currently already on study intervention(s).
5. Co-enrolment in another interventional trial (co-enrolment in an observational study is permitted).
6. Currently pregnant or breastfeeding.
7. The participant is currently enrolled in another clinical trial to treat neurocognitive symptoms in LC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Mean change in Modified Fatigue Impact Scale (MFIS) from baseline to three months | Three months
  This study will target detection of a change in the MFIS from baseline to three months
Mean change in the ratio of the Trail-Making Tests A & B in the TestMyBrain cognitive testing battery from baseline to three months. | Three months
  This test will target detection of a change in the ratio of the Trail-Making Tests A & B from baseline to three months

SECONDARY OUTCOMES:
Core Outcome Set - Symptoms | Three months
  Tracking of symptom trajectory from baseline to three months
Cardiovascular function | Three months
  Mean change in results of 6-minute walking test, to include symptoms and conditions
Respiratory function | Three months
  Mean change in results of 6-minute walking test, to include symptoms and conditions
Cognitive Function | Three months
  Measurement of mean change in cognition using the TestMyBrain assessment tool.
Memory | Three months
  Measurement of mean change in memory using the TestMyBrain assessment tool.
Concentration | Three months
  Measurement of mean change in concentration using the TestMyBrain assessment tool.
Conceptual Thinking | Three months
  Measurement of mean change in conceptual thinking using the TestMyBrain assessment tool.
Social Functioning | Three months
  Measurement of mean change in social functioning using the TestMyBrain assessment tool.
Mental Health Status - PHQ-9 | Three months
  Measurement of mean change in mental health status using the Patient Health Questionnaire (PHQ-9).
Mental Health Status - GAD-7 | Three months
  Measurement of mean change in mental health status using the General Anxiety Disorder Questionnaire (GAD-7).
Post-Exertional Malaise (PEM) Symptoms | Three months
  Measurement of changes in onset and triggers of PEM, symptoms, duration and recovery using the Post-Exertional Malaise questionnaire, adapted from De Paul's Symptom Questionnaire (PEM-DSQ).
Post-COVID-19 Functional Status (PCFS) Scale | Three months
  Measurement of changes in post-COVID functional status using the Post-COVID-19 Functional Status (PCFS) Scale.
Reintegration to Normal Living Index (RNLI) | Three months
  Measurement of changes in reintegration to normal social activities using the Reintegration to Normal Living Index (RNLI) assessment tool.
Health Related Quality of Life - SF-36 (v.1) | Three months
  Measurement of change in quality of life using the Quality of Life - SF-36 (v.1) assessment tool.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Richer, MD, MSc, Principal Investigator — University of Alberta
Locations (4):
- Canada (4):
  - University of Alberta Hospital, Kaye Edmonton Clinic, Edmonton, Alberta
  - University Health Network, Toronto, Ontario
  - Institut de recherches cliniques de Montréal, Montreal, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec